CLINICAL TRIAL: NCT06553521
Title: Universal Psychosocial Screening Using MyHEARTSMAP In Hospitalized Pediatric Patients: A Randomized Control Study
Brief Title: MyHEARTSMAP In-Patient Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Quynh Doan, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H21-01221
Record Dates: First submitted 2024-06-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Issue; Psychosocial Functioning
Keywords: screening tool; randomized control trial; psychosocial screening; in-patient; universal mental health screening; pediatrics; universal psychosocial screening; pediatric mental health; mental health screening; MyHEARTSMAP

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Other): In the MyHEARTSMAP intervention group, research assistants (RAs) help with the self-administered screening using a device. Validated for ages 10-17, both self-reporting and proxy-reporting are allowed.
  After self- and/or parent-reports, a MyHEARTSMAP report is auto-submitted to REDCap, with one printed copy for the patient chart. if there are any mental health concerns identified in MyHEARTSMAP report, they will be addressed by the treating teams. Respondents can receive reports via email, ensuring privacy and separate reports for parents and youth. Discussions with the treating team are encouraged. Severe safety concerns during ED screening prompt immediate contact with the treating team. The admitting service manages concerns in the care plan.
  Interventions: Other: MyHEARTSMAP Youth Self-assessment Tool (At Admission)
- Standard of care (delayed MyHEARTSMAP arm): (No Intervention): Participants receiving standard care will complete an initial data collection form for demographic and medical information. After hospital discharge, they'll get a link to complete MyHEARTSMAP. Reminder email will be sent if MyHEARTSMAP is not completed by days 3 and 7.
  Severe or acute safety concerns from MyHEARTSMAP trigger alerts, directing participants to crisis lines or EDs. RAs review daily for such concerns, contacting the research team for follow-up, led by a pediatric emergency physician.

INTERVENTIONS:
Other: MyHEARTSMAP Youth Self-assessment Tool (At Admission) — MyHEARTSMAP is a validated self-assessment tool for pediatric populations, demonstrating high sensitivity and specificity for identifying psychosocial concerns. Adapted from HEARTSMAP, it allows self- and proxy-reporting across 10 well-being domains, providing personalized recommendations. Currently, the clinician-reported HEARTSMAP is the standard of care at BC Children's Hospital ED for the initial assessment of youth with primary psychiatric concerns
  Arms: Intervention arm

SUMMARY:
Often, mental health (MH) conditions are under-identified in youth with chronic health conditions, which can lead to long-term health consequences and can impact their everyday lives. Hospitalized youth often experience higher MH burdens and tend to have fewer interactions with their primary healthcare providers upon discharge, leading to overall worse health outcomes. In-hospital treatment focuses on the acute physical condition relating to the hospitalization and often neglects the mental health aspect of the patients general health problems. The American Academy of Paediatrics has advocated for the universal use of MH screening tools to detect and facilitate management of youth with psychiatric illnesses; however, this has yet to be effectively implemented. Currently, the guidelines for screening of MH related concerns in hospitalized youth vary by treating specialties. The investigators believe that having a universal psychosocial screening using an online MH self-assessment tool, MyHEARTSMAP, in hospitalized youth will allow for early screening of MH conditions and can improve their holistic biopsychosocial care.

DETAILED DESCRIPTION:
Purpose/Objective: The goal of this project is to investigate if implementing universal psychosocial screening using the MyHEARTSMAP instrument in hospitalized pediatric patients admitted for non primary psychiatric concerns increase/affect their holistic biopsychosocial management.

Hypothesis/Justification: Mental health conditions represent an increasingly substantial burden of illness in the pediatric population. Especially among youth who are hospitalized or experiencing chronic illness, there is a disproportionate burden of mental health concerns. However, large proportion of children who screen positive for mental health concerns while in hospital have never been identified as having a mental health concern, or have received health or social services related to such concerns.

The American Academy of Paediatrics has advocated for the universal use of efficient, culturally sensitive, and age-appropriate mental health screening tools to detect and facilitate management of youth with psychiatric illnesses; however, this has yet to be effectively implemented. Currently, in Canada, anecdotal evidence suggests that the standard of care for screening mental health related concerns in hospitalized youth typically varies by treating specialty. The lack of a consistent, systematic approach to screening youth coupled with reduced screening among those with higher medical needs may result in vulnerable pediatric populations falling through gaps of care in medical systems. In order to address the issue of under-identification of mental health illness in youth requiring hospitalization, this study proposes to implement a universal mental health screening using an online self-assessment tool, MyHEARTSMAP, in hospitalized youth to allow for early screen of mental health conditions and to improve their holistic biopsychosocial care.

MyHEARTSMAP has been validated as a universal screening tool and, when compared to clinician reports, has high sensitivity and specificity to identify youth with psychosocial concerns that warrant further follow-up. Upon completion of the tool, MyHEARTSMAP produces triggered recommendations that are consistent with clinician assessment. This tool has been adapted from HEARTSMAP, a clinical assessment tool used by British Columbia (BC) Children's Hospital Paediatric ED clinicians for mental health assessment and management of youth presenting with mental health concerns. Designed for self-assessment and universal screening, MyHEARTSMAP allows children and their parents to efficiently self- and proxy-report across multiple domains of mental health. MyHEARTSMAP allows for the comprehensive evaluation of 10 areas of wellbeing that makeup the 'HEARTSMAP' acronym: Home, Education and activities, Alcohol and drugs, Relationships and bullying, Thoughts and anxiety, Safety, sexual health, Mood, Abuse, and Professional resources.

Study Design, Population and Setting: The investigators propose to conduct a prospective randomized controlled study to evaluate the impact of standardized psychosocial screening using MyHEARTSMAP upon admission to an in-patient ward, on the frequency of psychosocial intervention during the hospitalization or mental health resource referrals upon discharge.

Statistical Analysis: The investigators will use descriptive statistics to summarize our study population demographic distributions. Our primary objective of comparing the proportion of participants receiving psychosocial interventions as part of their in-patient care or at discharge will be analysed using a test of proportions. Our secondary and exploratory analyses will include: comparing the proportion of youth who receive psychosocial interventions or mental health resources during the three-month period following discharge. The investigators will additionally report why or why not resources were accessed in the community, including barriers reported. The investigators will use NVivo to analyze descriptive responses and code by theme to describe barriers to mental health resource access and include representative quotes.

Sample Size: The investigators know from previous studies that approximately 40% of youth who present to the ED will screen positive in at least one domain of HEARTSMAP with recommendations to follow-up with specific resources. The investigators presume that at least 80% of those will receive services within their hospital stay or referrals at the time of discharge, or 30% of participants randomized to screening with MyHEARTSMAP. Given these factors, to achieve a power of 80% and 95% confidence, to detect an absolute difference of 15% (or relative difference of 50%) in proportion of youth who receive psychosocial interventions between study arms, the investigators would need to recruit 135 participants per arm. Accounting for 30% attrition (25% in previous MyHEARTSMAP studies), a sample size of 175 per arm is required.

ELIGIBILITY:
Inclusion Criteria:

* Children and youth aged 7-17 years (and their guardians) from the emergency department (ED)
* Primary non-psychiatric concerns
* Admitted to the in-patient general pediatrics, cardiology, nephrology, neurology, endocrinology, gastroenterology, general surgery, urology, or orthopaedic surgery services OR from the surgical units if they have a pre-planned admission under general surgery, orthopaedic surgery, or urology for an elective surgery
* Use of translators in the ED or surgical units will be accessed as available (ED/surgical unit staff with shared language skills) to help include families with language barrier challenges.

Exclusion Criteria:

* Hospitalized with a mental health condition as the primary reason for their ED visit or surgery.
* Requiring a sustained level of critical care
* Aged <7 and >17 years at the time of ED presentation or surgery
* Previously enrolled in the study (ie. multiple admissions)
* No email and internet access (email and internet access is required in order to access MyHEARTSMAP if completing after discharged from hospital.)
* No mental capacity to read, understand and agree to the assent form.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 289 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Incorporation of mental health resources during in-patient stay | During admission period
  The investigators will report the proportion of youth who received MH resources/consultation during their in-patient stay comparing participants in their randomized intervention group.
Incorporation of MH resources on discharge planning | Time at which participant is discharged from hospital, could be up to approximately 6 weeks from date of randomization
  The investigators will compare the proportion of youth who received MH resources and recommendations for support on their discharge plans comparing participants in their randomized intervention group. The investigators will also assess whether the care team provided verbal consultation with patients/families at the time of discharge.

SECONDARY OUTCOMES:
Utilization of mental health resources following discharge | At 3 months following discharge
  At the 3-month follow-up, all participating families will receive, by email, a link to a survey to assess whether they have accessed any psychosocial resources or therapeutics since discharge. They will also be prompted to indicate what barriers prevented them from accessing care if it was so indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No